CLINICAL TRIAL: NCT02616588
Title: Vets Helping Vets Pilot Study
Acronym: VHV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-2137
Record Dates: First submitted 2015-11-20; First posted 2015-11-30 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Advanced Stage Cancer
Keywords: advanced stage cancer,; patient navigator,; social work
MeSH Terms: interventions — Social Work

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Arm (Experimental): All participants are enrolled into the intervention arm and receive the Veteran Patient Navigator and Social Work Intervention.
  Interventions: Behavioral: Veteran Patient Navigator and Social Work Intervention

INTERVENTIONS:
Behavioral: Veteran Patient Navigator and Social Work Intervention — Each study participant will receive a veteran patient navigator intervention which consists of five study visits consisting of advance care planning, pain/symptom management, and education about hospice and palliative care. When clinically indicated, patients will be referred to a social work intervention providing psychosocial care and support.

SUMMARY:
The overall goal of this study is to evaluate the feasibility of a veteran patient navigator and social work counseling intervention in veterans with advanced stage cancer at the Denver VA Medical Center. This is a tiered intervention: patients first receive the veteran patient navigator component of the intervention, and then if additional patient needs are present they receive the social work counseling component of the intervention. The overall intervention will help veterans communicate their care preferences with their providers.This is a study of behavioral and care strategy interventions and involves no investigational drugs or devices.

DETAILED DESCRIPTION:
Many patients with advanced cancer suffer from multiple symptoms including pain and fatigue and high rates of depression and anxiety. Many also experience end of life care that is inconsistent with their preferences.

Recent studies of palliative care find that symptoms, depression, and end of life care quality improved in patients with advanced cancer with multidisciplinary, specialist palliative care compared to usual care. However, these palliative care interventions are personnel-intensive and require multiple specialist providers. Because of the costs and limited availability of specialist palliative care providers, these interventions cannot be spread to the large population of patients with advanced cancer. Thus, there is a need for scalable interventions to improve symptoms, depression, and end of life care in this patient population.

Patient navigators, who often belong to the community they serve, have improved rates of cancer screening, follow up on abnormal diagnostic tests, and adherence to chemotherapy regimens. There has been increasing recognition that palliative care is an important part of patient navigation. However, to the best of our knowledge, there have been no studies outside our research program that have examined the effects of a peer navigation intervention to improve palliative care outcomes.

While patient navigators hold promise for improving outcomes in patients with advanced cancer, both psychosocial care needs and documenting future care preferences and goals may be complex. Therefore, the proposed intervention will supplement veteran patient navigators with a social work psychosocial intervention. The goal of the proposed study is to evaluate the feasibility of a stepped care intervention including a veteran patient navigator and social worker.

ELIGIBILITY:
Inclusion Criteria:

* Adult (over 18 years of age)
* Patient has an oncology provider within the VA ECHCS
* English is patient's primary language
* Has a reliable telephone
* Diagnosis of cancer deemed as incurable by oncology provider
* Oncology provider answers "no" to the question, "Would you be surprised if this patient dies in the next year?"

Exclusion Criteria:

* Already receiving specialist palliative care or receiving hospice care

Ages: 18 Years to 108 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-02; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Aim 1A. Examine intervention feasibility. | 1 year
  The intervention will be feasible if:
  A. The participation rate is above 40% and the retention rate is above 60%.
Aim 1B. Examine intervention feasibility. | 1 year
  The intervention will be feasible if:
  B. Oncology providers and patient participants find the intervention acceptable as defined by mean ratings of above "somewhat" useful/helpful/satisfied (i.e., above 3 on a 1 to 5 Likert scale, where 5 is "extremely" and 1 is "not at all."
Aim 1C. Examine intervention feasibility. | 1 year
  The intervention will be feasible if:
  C. There is less than 10% missing data on patient-reported survey measures.

SECONDARY OUTCOMES:
Aim 2A. aTrack intervention process in order to improve the intervention | 1 year
  A. Determine patient flow through the intervention and adherence to the study protocol by tracking:
  a. number of visits
Aim 2Ab. Track intervention process in order to improve the intervention | 1 year
  A. Determine patient flow through the intervention and adherence to the study protocol by tracking:
  b. visit length
Aim 2Ac. Track intervention process in order to improve the intervention | 1 year
  A. Determine patient flow through the intervention and adherence to the study protocol by tracking:
  c problem addressed
Aim 2Ad. Track intervention process in order to improve the intervention | 1 year
  A. Determine patient flow through the intervention and adherence to the study protocol by tracking:
  d. who is seen by the social worker and why
Aim 2Ae. Track intervention process in order to improve the intervention | 1 year
  A. Determine patient flow through the intervention and adherence to the study protocol by tracking:
  e. adherence to the study protocol
Aim 2B. Track intervention process in order to improve the intervention | 1 year
  B. Understand patient and oncology provider reactions through qualitative interviews to the intervention to inform how to improve feasibility or helpfulness.

CONTACTS AND LOCATIONS:
Overall Officials: David Bekelman, MPH, MD, Principal Investigator — Eastern Colorado Health Care System, Department of Veterans Affairs, Denver, CO

REFERENCES:
- [Background] Arrieta O, Angulo LP, Nunez-Valencia C, Dorantes-Gallareta Y, Macedo EO, Martinez-Lopez D, Alvarado S, Corona-Cruz JF, Onate-Ocana LF. Association of depression and anxiety on quality of life, treatment adherence, and prognosis in patients with advanced non-small cell lung cancer. Ann Surg Oncol. 2013 Jun;20(6):1941-8. doi: 10.1245/s10434-012-2793-5. Epub 2012 Dec 22. PMID 23263699
- [Background] Mack JW, Weeks JC, Wright AA, Block SD, Prigerson HG. End-of-life discussions, goal attainment, and distress at the end of life: predictors and outcomes of receipt of care consistent with preferences. J Clin Oncol. 2010 Mar 1;28(7):1203-8. doi: 10.1200/JCO.2009.25.4672. Epub 2010 Feb 1. PMID 20124172
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Zimmermann C, Swami N, Krzyzanowska M, Hannon B, Leighl N, Oza A, Moore M, Rydall A, Rodin G, Tannock I, Donner A, Lo C. Early palliative care for patients with advanced cancer: a cluster-randomised controlled trial. Lancet. 2014 May 17;383(9930):1721-30. doi: 10.1016/S0140-6736(13)62416-2. Epub 2014 Feb 19. PMID 24559581
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Block SD, Billings JA. A need for scalable outpatient palliative care interventions. Lancet. 2014 May 17;383(9930):1699-700. doi: 10.1016/S0140-6736(13)62676-8. Epub 2014 Feb 19. No abstract available. PMID 24559580
- [Background] Freeman HP. Patient navigation: a community based strategy to reduce cancer disparities. J Urban Health. 2006 Mar;83(2):139-41. doi: 10.1007/s11524-006-9030-0. No abstract available. PMID 16736361
- [Background] Freeman HP, Muth BJ, Kerner JF. Expanding access to cancer screening and clinical follow-up among the medically underserved. Cancer Pract. 1995 Jan-Feb;3(1):19-30. PMID 7704057
- [Background] Steinberg ML, Fremont A, Khan DC, Huang D, Knapp H, Karaman D, Forge N, Andre K, Chaiken LM, Streeter OE Jr. Lay patient navigator program implementation for equal access to cancer care and clinical trials: essential steps and initial challenges. Cancer. 2006 Dec 1;107(11):2669-77. doi: 10.1002/cncr.22319. PMID 17078056
- [Background] Wells KJ, Battaglia TA, Dudley DJ, Garcia R, Greene A, Calhoun E, Mandelblatt JS, Paskett ED, Raich PC; Patient Navigation Research Program. Patient navigation: state of the art or is it science? Cancer. 2008 Oct 15;113(8):1999-2010. doi: 10.1002/cncr.23815. PMID 18780320
- [Background] Calhoun EA, Whitley EM, Esparza A, Ness E, Greene A, Garcia R, Valverde PA. A national patient navigator training program. Health Promot Pract. 2010 Mar;11(2):205-15. doi: 10.1177/1524839908323521. Epub 2008 Dec 30. PMID 19116415
- [Background] Freeman HP, Chu KC. Determinants of cancer disparities: barriers to cancer screening, diagnosis, and treatment. Surg Oncol Clin N Am. 2005 Oct;14(4):655-69, v. doi: 10.1016/j.soc.2005.06.002. PMID 16226685
- [Background] Freeman HP. Patient navigation: a community centered approach to reducing cancer mortality. J Cancer Educ. 2006 Spring;21(1 Suppl):S11-4. doi: 10.1207/s15430154jce2101s_4. PMID 17020496
- [Background] Fischer SM, Cervantes L, Fink RM, Kutner JS. Apoyo con Carino: a pilot randomized controlled trial of a patient navigator intervention to improve palliative care outcomes for Latinos with serious illness. J Pain Symptom Manage. 2015 Apr;49(4):657-65. doi: 10.1016/j.jpainsymman.2014.08.011. Epub 2014 Sep 18. PMID 25240788